CLINICAL TRIAL: NCT01325753
Title: A Pilot Study of Cryoablation for Patients With Oligometastatic Cancer Involving the Lung
Brief Title: Cryotherapy in Treating Patients With Lung Cancer That Has Spread to the Other Lung or Parts of the Body
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00015085; NCI-2011-00319 (Registry Identifier: CTRP); CCCWFU 62210 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Advanced Malignant Mesothelioma; Extensive Stage Small Cell Lung Cancer; Lung Metastases; Recurrent Malignant Mesothelioma; Recurrent Non-small Cell Lung Cancer; Recurrent Small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Mesothelioma, Malignant; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (cryoablation) (Experimental): Patients undergo CT-guided CA.
  Interventions: Procedure: cryotherapy; Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: cryotherapy — Undergo CT-guided CA
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This pilot clinical trial studies the side effects of cryotherapy (cryoablation [CA]) in treating patients with lung cancer. Cryotherapy kills cancer cells by freezing them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the initial safety of the CA for lung tumors less than or equal to 3.5 cm in size including acute toxicity (30 days).

SECONDARY OBJECTIVES:

I. Estimate local control.

II. To assess physical function for this cohort of patients.

III. To evaluate the impact of treatment on generic and disease-specific quality of life.

IV. To obtain pilot data useful for the design of a subsequent phase II or randomized phase II trial.

V. Evaluate changes in pulmonary function at 3 months.

OUTLINE:

Patients undergo computed tomography (CT)-guided CA

After completion of study treatment, patients are followed up at 1 week and 1, 3, 6, 12, 24, 36, 48, and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Joint Committee on Cancer (AJCC) seventh edition metastatic carcinoma or sarcoma involving the lungs or pleura.
* Pathologic diagnosis of stage 4 cancer prior to enrollment by biopsy or on imaging with known (biopsied) primary disease
* The target lesion is determined (by CT or magnetic resonance imaging [MRI] images) to be in a location where cryoablation is technically achievable based on the proximity of adjacent organs and structures
* Maximum number of lesions per patient will be 5 total (a maximum of 3 on either the right or left side and 2 lesions on the respective contralateral side)
* Of these, any lesion not treated with cryoablation will be planned to be treated with radiotherapy or radiofrequency ablation, such that all known active pulmonary disease is planned to be treated with a definitive local therapy
* If treatment of both lungs is to occur by cryoablation, these treatments must be separated by at least one week
* The lesion(s) treated with cryoablation may be intrapulmonary or pleural and must be =< 3.5 cm in greatest dimension
* All patients are required to have been evaluated either in consultation with a radiation oncologist or at least in a multi-disciplinary tumor conference to ensure that all local therapy options are appropriately considered for each patient
* Performance Status 0-2 (Eastern Cooperative Oncology Group [ECOG]); Karnofsky Performance Scale >= 60
* Life expectancy > 3 months
* Clinically suitable for cryoablation procedure as determined by the treating physician
* Platelet count > 50,000/mm^3 within 60 days prior to study registration
* International normalized ratio (INR) < 1.5 within 60 days prior to study registration
* Absolute neutrophil count (ANC) < 1000 within 21 days prior to study registration
* A signed study specific consent form is required

Exclusion Criteria:

* Primary lung cancer
* Unable to lie flat or has respiratory distress at rest
* Uncontrolled coagulopathy or bleeding disorders
* Evidence of active systemic, pulmonary, or pericardial infection
* Pregnant, nursing or wishes to become pregnant during the study
* Debilitating medical or psychiatric illness that would preclude giving informed consent or receiving optimal treatment or follow up
* Currently participating in other experimental studies that could affect the primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Safety of interventional cryoablation to the lung | 6 months
  Unexpected toxiticities or Grade 4 or 5 toxicities will be recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Local control measured by imaging | At 1 year
  Measure definitions:
  * Complete Response(tumor disappearance or less than 25% of original size)
  * Partial Response (greater than 30% decrease in the sum of the largest diameter of all targeted tumors)
  * stable Disease (less than 30% decrease in the sum of the largest diameter of all targeted tumors)
  * Local Failure (greater than 20% increase in the sum of the largest diameter of all targeted tumors)
  * Distant Failure (the appearance of distant cancer deposits consistent with metastatic spread of cancer outside the intended treatment area)
Changes in Physical function and quality of life | approximately 60 months
  Measured by ECOG and KPS performance status, the Short Form - 12v2 questionnarie and shory physical performance battery
Changes in pulmonary function | At 3 months
  Measure by pulmonary function test
Obtain pilot data useful for the design of a subsequent phase II or randomized phase II trial | approximately 60 months

CONTACTS AND LOCATIONS:
Overall Officials: James Urbanic, Principal Investigator — Wake Forest University Health Sciences